CLINICAL TRIAL: NCT02988570
Title: Study on the Phenotype of Language in Preterm Born Children at 5 Years of Age
Acronym: EPILANG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/338/HP
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Preterm Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- children born very preterm (Experimental): A computer-evaluation of the language will be done for children born very preterm preterm in 2011 in the region of Haute-Normandie in France
  Interventions: Behavioral: computer-evaluation of the language

INTERVENTIONS:
Behavioral: computer-evaluation of the language — A computer-evaluation of the language will be done for children born very preterm preterm in 2011 in the region of Haute-Normandie in France

SUMMARY:
In recent years, several studies confirm that some of preterm children have language developmental disabilities, in production, in comprehension, or in written language. These language impairments lead to learning disabilities. There are, however, contradictions concerning the origin and nature of language dysfunctions. Some studies find lexical disorders (number of words used by the child), others preferentially phonological disorders (sounds used in the language), others also disorders of the morphosyntaxe (organization of the sentences) and fragilities that affect pragmatics (understanding situations).

The computer-evaluation of the language is carried out at five and a half year coupled with the medical and neuropsychological examinations. The language assessment lasts 30 to 45 minutes per child. It is carried out using a laptop computer that allows the submission of stimuli and recording of the child's responses. The language evaluation scale is the battery CléA (Pasquet F et al, 2014), standardized reference tool for the realization of a language evaluation. The assessment includes three tests: comprehension of words and phrases, production of words and phrases, and judgment of sentences. Each time, the child sees images and hears words or phrases. Sometimes he has to say what he sees on the computer screen.

As usual, a speech-language assessment is not carried out, routinely, at the age of 5 years in the context of the follow-up of children born very preterm.

The evaluation proposed to the child in this research will be carried out at a significant period of development, before writing. This assessment will not only assess the structure of the child's language, but also determine if there are possible difficulties in learning to read and write.

The expected benefits for the health of the children included in the trial therefore concern the detection or characterization of any developmental fragilities affecting the language. These screenings or characterizations will make it possible to advocate a speech rehabilitation if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Children born very preterm in 2011 in the region of Haute-Normandie in France

Exclusion Criteria:

* None

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of comprehension of words and phrases level | Day 1
  A computer-based language evaluation battery (Cléa) comprising standardized test to evaluate comprehension of words and phrases will be used.

SECONDARY OUTCOMES:
Evaluation of production of words and phrases level | Day 1
  A computer-based language evaluation battery (Cléa) comprising standardized test to evaluate production of words and phrases level will be used.
Evaluation of judgment of sentences level | Day 1
  A computer-based language evaluation battery (Cléa) comprising standardized test to evaluate judgment of sentences level will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane MARRET, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No